CLINICAL TRIAL: NCT07277127
Title: Effect of Percutaneous Electrolysis Combined With Exercise on Pain and Function in Chronic Lateral Epicondylitis: A Randomized Controlled Trial
Brief Title: Effect of Percutaneous Electrolysis Combined With Exercise on Pain and Function in Chronic Lateral Epicondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sivas State Hospital (Other)
Responsible Party: Principal Investigator, Serkan Polat, MD, Sivas State Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPTE-001-S
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): Participants perform a 2-week exercise program including stretching and eccentric strengthening exercises for the wrist extensor and forearm muscles.
  Interventions: Other: Exercise
- Percutaneous Electrolysis plus Exercise (Experimental): Participants receive the same 2-week exercise program as the control group plus three sessions of ultrasound-guided percutaneous electrolysis applied to the extensor carpi radialis brevis tendon insertion at the lateral epicondyle on days 1, 8, and 14.
  Interventions: Other: Exercise; Device: Percutaneous Electrolysis

INTERVENTIONS:
Other: Exercise — 2-week exercise program with stretching and eccentric strengthening for wrist extensors and forearm muscles.
Device: Percutaneous Electrolysis — Participants receive the same 2-week exercise program as the control group plus three sessions of ultrasound-guided percutaneous electrolysis applied to the extensor carpi radialis brevis tendon insertion at the lateral epicondyle on days 1, 8, and 14.
  Arms: Percutaneous Electrolysis plus Exercise

SUMMARY:
The aim of this randomized controlled trial is to compare the effects of percutaneous electrolysis combined with exercise versus exercise alone on pain and function in patients with chronic lateral epicondylitis. Participants will be randomly allocated into two parallel groups. The control group will receive a 2-week exercise program including stretching and eccentric strengthening exercises for the wrist extensor and forearm muscles. The experimental group will receive the same exercise program plus three sessions of ultrasound-guided percutaneous electrolysis applied to the extensor carpi radialis brevis tendon insertion at the lateral epicondyle (on days 1, 8, and 14). Clinical outcomes will be assessed using a 10-cm Visual Analog Scale (VAS) for pain intensity, pressure pain threshold over the common extensor tendon measured with a handheld algometer, the Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire for pain and functional disability, and the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire for upper limb function. Assessments will be performed at baseline, and then at 1 week, 1 month, and 3 months after the end of the 2-week treatment period. The study aims to determine whether adding percutaneous electrolysis to an exercise program provides greater improvement in pain and functional status than exercise alone in patients with chronic lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Clinically and MRI-confirmed diagnosis of chronic lateral epicondylitis (symptoms ≥ 3 months)
* Ability and willingness to comply with the treatment protocol and follow-up schedule

Exclusion Criteria:

* Previous elbow surgery or fracture in the affected limb
* Local corticosteroid injection or other invasive treatment in the past 3 months
* Cervical radiculopathy, systemic rheumatic disease, or other neurological disorders affecting the upper limb
* Presence of a cardiac pacemaker or diagnosis of epilepsy
* Pregnancy or breastfeeding
* Serious bleeding disorder (coagulopathy) or current anticoagulant therapy
* Inability to follow the exercise protocol or attend follow-up visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity (VAS) | Baseline, 1 week post-treatment, 1 month, 3 months
  Pain intensity will be measured using a 10-cm Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Change in Pressure Pain Threshold (Algometry) | Baseline, 1 week post-treatment, 1 month, 3 months
  Pressure pain threshold over the common extensor tendon will be measured using a handheld algometer.
Change in Functional Status (PRTEE Score) | Baseline, 1 week post-treatment, 1 month, 3 months
  Functional disability and pain will be assessed using the Patient-Rated Tennis Elbow Evaluation (PRTEE).
Change in Upper Limb Function (QuickDASH) | Baseline, 1 week post-treatment, 1 month, 3 months
  Upper limb disability will be evaluated using the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas State Hospital, Sivas, Turkey (Türkiye)